CLINICAL TRIAL: NCT04329039
Title: Randomized Control Trial Comparing Somatostatin Analogues With Perioperative Antibiotics Versus Prolonged Antibiotics
Brief Title: Somatostatin Analogues With Perioperative Antibiotics Versus Prolonged Antibiotics
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18-010128; NCI-2022-11062 (Registry Identifier: NCI)
Record Dates: First submitted 2020-03-30; First posted 2020-04-01 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Pancreatic Diseases
MeSH Terms: conditions — Pancreatic Diseases | interventions — Somatostatin

STUDY DESIGN:
Intervention Model Description: Randomized control trial comparing somatostatin analogues with perioperative antibiotics versus prolonged antibiotics
Who Masked: Participant
Masking Description: Patients will be randomized on a 1:1 ratio to either somatostatin analogues with perioperative antibiotics vs. placebo with perioperative antibiotics
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Active Comparator): Active somatostatin analogue combined with perioperative antibiotics
  Interventions: Drug: Somatostatin analog
- Group 2 (Placebo Comparator): Placebo combined with perioperative antibiotics
  Interventions: Drug: Somatostatin analog

INTERVENTIONS:
Drug: Somatostatin analog — Somatostatin analog plus perioperative antibiotics Placebo plus perioperative antibiotics
  Other Names: Arm A

SUMMARY:
Researchers are trying to determine how the length of antibiotic treatment in addition to octreotide after pancreatic surgery affects the amount of time subjects are hospitalized as well as how many subjects develop pancreatic fistulas.

ELIGIBILITY:
Inclusion Criteria

* Patients undergoing a Whipple procedure for various diagnoses (neuroendocrine tumors, adenocarcinoma, benign cystic neoplasms, duodenal and ampullary malignancies, etc) who are deemed intermediate-high risk as per our institutional protocol as shown above.
* Patients > 18 years of age

Exclusion Criteria

* Negligible and low risk patients
* All patients undergoing arterial resection.
* Age <18 years
* Currently pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2020-11-17 (Actual); Primary Completion 2025-02-07 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
This study aims to determine whether duration of antibiotic therapy coupled with octreotide leads to reduction of the severity or occurrence of pancreatic fistula. | During operative time plus 2 to 5 days post op
  To compare the active study medication with placebo to see if there is a reduction in the active drug arm in occurrence or pancreatic fistula

CONTACTS AND LOCATIONS:
Overall Officials: Michael L Kendrick, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials